CLINICAL TRIAL: NCT07248293
Title: "Investigation of the Effect of Income Level in Older Adults: A Randomized Controlled Trial"
Brief Title: "Income Level and Its Effect in Older Adults"
Status: Completed | Type: Observational
Sponsor: Begüm AKAR (Other)
Responsible Party: Sponsor-Investigator, Begüm AKAR, Principal investigator, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: Pamukkale U
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Older Adults (65 Years and Older)
Keywords: older adults
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- minimum wage: Minimum Wage Group:
  The elderly in this group consist of older adults earning a minimum wage.
  Interventions: Other: Behavioral Treatment; Behavioral: behavioral
- above minimum wage group: Above Minimum Wage Group:
  The elderly in this group consist of older adults whose income levels are above the minimum wage threshold.
  Interventions: Other: Behavioral Treatment; Behavioral: behavioral

INTERVENTIONS:
Other: Behavioral Treatment — What makes this study different is that participants are categorized according to income levels, and detailed analyses are conducted between the subgroups.
Behavioral: behavioral — The difference between this study and other studies is that in this study, the elderly are categorized according to their income levels.

SUMMARY:
The aim of this study was to examine the effect of income level on cognitive function, pain, balance, lower extremity performance, gait, occupational competence, depression, and health-promoting behaviors in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years of age or older
* Volunteering to participate in the study
* Elderly individuals scoring 6 or higher on the Hodkinson Mental Test

Exclusion Criteria:

* Elderly individuals who cannot communicate due to conditions such as Alzheimer's disease, dementia, or psychosis
* Having another chronic disease that may cause pain (rheumatic diseases, hemiplegia, multiple sclerosis, diabetes, etc.)
* Having a neurological disease (hemiplegia, Parkinson's disease, multiple sclerosis, vertigo, epilepsy, etc.)
* Being blind
* Having orthopedic, neurological, or mental disabilities

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: elderly
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE): | 10 minutes
  Mini-Mental State Examination (MMSE):
  The Mini-Mental State Examination is a scale used to assess individuals' cognitive status. It evaluates attention, orientation, memory, the ability to follow verbal and written commands, spontaneous writing, and copying complex drawings. The total score is 30, with a cutoff point of 24; scores below 24 indicate cognitive impairment. The Turkish validity and reliability study was conducted by Güngen et al. in 2002
Hodkinson mental test | 10 minutes
  The Hodkinson Mental Test was developed by H.M. Hodkinson in 1972 and is used to assess cognitive functions in older adults. The test consists of 10 questions in total, with each correct answer worth 1 point. Scores below 7 indicate cognitive impairment. The test can be completed in less than 5 minutes and is a short, easy-to-administer tool that does not include culturally specific questions .
Dominant Side Single-Leg Stance Test | 1 minutes
  Dominant Side Single-Leg Stance Test:
  In this test, if the participant uses a walking aid, timing starts when they lift their dominant leg and release the aid; if not, timing begins when the dominant leg is lifted. The test ends when the foot touches the ground. If the participant can balance for more than 30 seconds, the test is completed. The duration is recorded in seconds. A result of less than 10 seconds indicates balance impairment, and less than 5 seconds indicates a risk of falling (17).
Sit-to-Stand Test | 2 minutes
  Sit-to-Stand Test:
  The participant, seated on a standard 43 cm-high chair with arms crossed over the shoulders, is asked to stand up and sit down as quickly as possible for 30 seconds. The number of full stands completed is recorded.
Modified Gait Efficacy Scale (MGES): | 3 minutes
  Modified Gait Efficacy Scale (MGES):
  The Modified Gait Efficacy Scale (MGES) is an adaptation of the original Gait Efficacy Scale (GES) used to assess an individual's confidence in walking safely and effectively. The MGES includes several questions measuring participants' confidence in various walking activities. These questions are typically answered on a Likert-type scale (e.g., 0 to 10), where 0 represents the lowest confidence and 10 represents the highest confidence (26).

SECONDARY OUTCOMES:
Geriatric Pain Scale | 5 minutes
  The Geriatric Pain Scale, developed by Ferrell BA and colleagues in 2000, is a 24-item multidimensional scale. It assesses five dimensions: pain-related withdrawal (items 6, 17, 18, 19, 20, 21, 24), pain intensity (items 1, 2, 3, 4, 5, 22, 23), pain with movement (items 9, 10, 11, 12), pain during strenuous activities (items 8, 13, 14), and pain during other activities (items 7, 15, 16, 17, 22). Twenty-two items are scored as "Yes" or "No," and 2 items are scored on a 0-10 scale. Total scores range from 0 to 100, with 0-30 indicating mild pain, 30-69 moderate pain, and 70 or above severe pain (31). The Turkish validity and reliability study was conducted by Dursun and Bektas (2017). The Cronbach's alpha for the entire scale was 0.85, with subscale alpha values ranging from 0.67 to 0.93 (19).
Yesavage Geriatric Depression Scale (GDS) - Short Form: | 10 minutes
  Yesavage Geriatric Depression Scale (GDS) - Short Form:
  The Yesavage Geriatric Depression Scale, developed in 1983, assesses depressive mood in older adults and is self-reported. The 15-item short form, validated in Turkish, scores depression-related items as 1 and non-depression items as 0, with five items reverse-scored (items 1, 5, 7, 11, 13). Scores range from 0 to 15, with higher scores indicating greater depressive symptoms. The cutoff point is 5. The scale has high internal consistency, with a Cronbach's alpha of 0.92.
Occupational Self Assessment (OSA) Scale: | 5 minutes
  The Occupational Self Assessment (OSA) Version 2.2 was used to evaluate individuals' occupational competence. Participants rate how well they perform 21 activities on a scale from 1 (I have a lot of difficulty doing this) to 4 (I do this extremely well) and the importance of these activities from 1 (Not important to me) to 4 (Extremely important to me). After answering the competence (Step 1) and value (Step 2) questions, participants select the areas they most want to change (Step 3) (27,28).

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Pamukkale, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No